CLINICAL TRIAL: NCT01710215
Title: Parkland-UT Southwestern PROSPR Center: Colon Cancer Screening in a Safety Net: Comparative Effectiveness of FIT, Colonoscopy, & Usual Care Screening Strategies
Brief Title: Comparative Effectiveness of FIT, Colonoscopy, & Usual Care Screening Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Parkland Health and Hospital System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 102011-069; 1U54CA163308-01 (NIH); NCT03404973 (obsolete NCT alias)
Record Dates: First submitted 2012-10-05; First posted 2012-10-19 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Neoplasms; Colorectal Cancer; Colon Cancer; Mass Screening; Health Services Research; Comparative Effectiveness Research
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): * No outreach mailed invitations.
  * Ordering of colonoscopy or FIT for screening at the discretion of the primary provider.
  * Follow up of abnormal tests and results reporting to the patient at the discretion of primary and specialty providers.
- FIT Screening Strategy (Experimental): * Mailed outreach invitation to complete FIT, including a test kit (1-sample FIT, simplified instructions on how to perform the test, and return mailer with prepaid postage).
  * Two "live" phone reminders from project staff 2 to 3 weeks after the invitation to encourage screening completion.
  * Centralized processes to promote guideline-based follow up.
  Interventions: Other: FIT Screening Strategy
- Colon Screening Strategy (Experimental): * Mailed outreach invitation to complete a colonoscopy, including a number to call to schedule a colonoscopy.
  * Two "live" phone call reminders from project staff 2 to 3 weeks after the mailed invitation to encourage screening completion.
  * Centralized processes to promote guideline-based follow up.
  Interventions: Other: Colon Screening Strategy

INTERVENTIONS:
Other: FIT Screening Strategy — * Mailed outreach invitation to complete FIT, including a test kit (1-sample FIT, simplified instructions on how to perform the test, and return mailer with prepaid postage).
  * Two "live" phone reminders from project staff 2 to 3 weeks after the invitation to encourage screening completion.
  * Centralized processes to promote guideline-based follow up.
  Arms: FIT Screening Strategy
Other: Colon Screening Strategy — * Mailed outreach invitation to complete a colonoscopy, including a number to call to schedule a colonoscopy.
  * Two "live" phone call reminders from project staff 2 to 3 weeks after the mailed invitation to encourage screening completion.
  * Centralized processes to promote guideline-based follow up.
  Arms: Colon Screening Strategy

SUMMARY:
Colorectal cancer (CRC) is the 2nd leading cause of cancer death in the US, though CRC death can be reduced by screening. However, there is uncertainty as to which screening strategy is most clinically and cost-effective from a population perspective where the aim is to optimize completion of the entire screening process continuum. Modeling studies suggest benefits and harms of colonoscopy and stool blood test strategies are similar, but generally assume 100% participation and subsequent clinically appropriate follow up--something never achieved in clinical practice. Comparative effectiveness studies of testing strategies, including comparisons of specific tests and approaches to optimizing effective test use, are necessary. Safety-net health systems care for populations at increased risk for adverse CRC outcomes, such as the uninsured and minorities, and have more limited resources. Therefore, safety-nets must resolve the uncertainty regarding the most effective screening strategy. The investigators will conduct a system-level, randomized comparative effectiveness trial of the benefits, harms, and costs of 3 screening strategies over 3 years, among 6000 patients age 50-64 years, who are not up-to-date with CRC screening, served by a large safety net health system. The three strategies studied will be: 1) Fecal immunochemical testing, with annual mailed invitation outreach (including a test kit), and a centralized process to promote participation and complete clinical follow up (FIT); 2) Colonoscopy, with annual mailed invitation outreach, and a centralized process to promote participation and complete clinical follow up (Colo); 3) Usual Care, with no mailed invitation outreach, and screening offered at primary care visits. The primary measure of benefit will be an outcome measure that summarizes patient-specific effective screening successes. The primary measure of harm will be screening non-participation. The primary measure of cost will be cost per-patient effectively screened. Our specific aims are to: 1) Compare benefits, harms, and costs of a FIT strategy versus a Colo strategy for CRC screening among patients not up-to-date with screening, and 2) Compare benefits, harms, and costs of a) the FIT strategy vs. Usual Care and b) the Colo strategy vs. Usual Care for CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 50-64 years
* Seen one or more times at a Parkland primary care clinic within one year (Index Year)
* Participants in Parkland's medical assistance program for the uninsured (Parkland Health Plus)
* All races and ethnicities

Exclusion Criteria:

* Up-to-date with CRC screening, defined by:

  1. Colonoscopy in the last 10 years
  2. Sigmoidoscopy in the last 5 years
  3. Stool blood test (FIT) in the last year
* Prior history of CRC, total colectomy, inflammatory bowel disease, or colon polyps
* Address or phone number not on file
* Incarcerated

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5999 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Benefit: Proportion of patients achieving one of the effective screening "successes." | All outcomes will be adjudicated within 3 years.
  The primary benefit measure will be defined by the proportion of patients achieving an effective screening "success" defined as:
  * Invited to colonoscopy (i.e. colo), responded to invite, determined to be too sick to scope by phone triage and clinical review
  * Screening colo completed, no cancer detected
  * Screening colo completed, cancer detected, 1st cancer treatment consultation visit completed
  * FIT screening completed, test normal, FIT repeated annually for 2 years
  * FIT screening completed, test abnormal, failed phone triage for direct scheduling for colo, and after GI clinic visit, determined to be too sick to scope
  * FIT screening completed, test abnormal, failed phone triage and clinical review, GI clinic visit, determined to be scopable, colo completed
  * FIT screening completed, test abnormal, colo completed, no cancer detected
  * FIT screening completed, test abnormal, colo completed, cancer detected, 1st cancer treatment consultation visit completed
Harm: Rate of screening non-participation. | All outcomes will be adjudicated within 3 years.
  The primary measure of harms will be the rate of non-screening because initial test completion is a basic prerequisite for prevention of adverse CRC outcomes by a screening process. It is a readily measurable, basic quality assessment. Processes associated with high rates of non-screening would be expected to result in poor long term CRC outcomes.
Cost: Cost per-patient effectively screened. | All outcomes will be adjudicated within 3 years.
  The primary measure of costs will be the cost per-patient effectively screened from the health system perspective, with effective screening defined by the proportion of patients achieving an effective screening "success." Follow up time for cost-assessment will start at randomization and end either when a patient reaches an effective screening "success" endpoint, or at the end of the three year-follow up time. This outcome addresses a practical question most health systems will have in assessing our screening strategy: What is the strategy specific cost per-patient effectively screened?

SECONDARY OUTCOMES:
Benefit: Number of CRCs, advanced adenomas, and adenomas detected. | All outcomes will be adjudicated within 3 years.
  Number of CRCs, advanced adenomas, and adenomas detected.
Benefit: Number of patients screened. | All outcomes will be adjudicated within 3 years.
  Number of patients screened, defined by the proportion of patients completing one time FIT or colonoscopy.
Harm: Number of CRCs diagnosed based on symptoms/signs rather than screening. | All outcomes will be adjudicated within 3 years.
  Number of CRCs diagnosed based on symptoms/signs rather than screening.
Harm: Ineffective screening. | All outcomes will be adjudicated within 3 years.
  Not achieving an effective screening "success." See definition of effective screening "successes" above.
Harm: Post-colonoscopy bleeding or perforation. | All outcomes will be adjudicated within 3 years.
  Post-colonoscopy bleeding or perforation.
Harm: Failed colonoscopy due to incomplete bowel prep or inability to reach cecum. | All outcomes will be adjudicated within 3 years.
  Failed colonoscopy due to incomplete bowel prep or inability to reach cecum.
Cost: Cost per patient screened. | All outcomes will be adjudicated within 3 years.
  Cost per patient screened.
Cost: Incremental costs for the FIT and Colo strategies relative to the Usual Care strategy. | All outcomes will be adjudicated within 3 years.
  Incremental costs for the FIT and Colo strategies relative to the Usual Care strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singal, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

REFERENCES:
- [Derived] Singal AG, Gupta S, Skinner CS, Ahn C, Santini NO, Agrawal D, Mayorga CA, Murphy C, Tiro JA, McCallister K, Sanders JM, Bishop WP, Loewen AC, Halm EA. Effect of Colonoscopy Outreach vs Fecal Immunochemical Test Outreach on Colorectal Cancer Screening Completion: A Randomized Clinical Trial. JAMA. 2017 Sep 5;318(9):806-815. doi: 10.1001/jama.2017.11389. PMID 28873161